CLINICAL TRIAL: NCT06707870
Title: Compare the Effectiveness of Cervical Retraction Exercise and Facet Oscillatory Mobilization in Improving Pain, Ranges and Disability in Patients With Chronic Mechanical Neck Pain.
Brief Title: Comparison of Cervical Retraction Exercise and Facet Oscillatory Mobilization in Chronic Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Riphah/RCRAHS/REC/MS-PT/01931
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Chronic Neck Pain
Keywords: Chronic neck pain; Facet oscillatory mobilization; Cervical retraction exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cervical retraction exercise (Experimental): Cervical retraction exercise
  Interventions: Other: Cervical retraction exercise
- Facet oscillatory mobilization (Experimental): Facet oscillatory mobilization
  Interventions: Other: Facet oscillatory mobilization

INTERVENTIONS:
Other: Cervical retraction exercise — Neck retraction exercises are performed on patients either in sitting or standing in an upright position while pushing their chin backward and simultaneously raising their head within the pain-free range (3 seconds hold)of 10 repetitions in each session at sitting position. Conventional treatment (TENS (2 to 10 Hz),10 mints, Heating pad, stretching of tight muscles Trapezius and SCM)should be included.
  The patients will received 20-30-minute sessions on 3 alternate days for two consecutive weeks, making it a total of 6 sessions. Patients were advised to revisit after 4 weeks (1 month from the baseline) for follow-up.
  Arms: Cervical retraction exercise
Other: Facet oscillatory mobilization — Facet joint oscillatory mobilization on the cervical spine C2-C7(6 to 10 repetitions in each session) in the sitting position.
  Conventional treatment (TENS (2 to 10 Hz) 10 mints, Heating pad, stretching of tight muscles Trapezius and SCM) should be included.
  The patients will received 20-30-minute sessions on 3 alternate days for two consecutive weeks, making it a total of 6 sessions. Patients were advised to revisit after 4 weeks (1 month from the baseline) for follow-up.
  Arms: Facet oscillatory mobilization

SUMMARY:
To compare the effects of Cervical Retraction Exercise and Facet Oscillatory Mobilization in chronic Mechanical Neck pain.

To compare the effects of Cervical Retraction Exercise and Facet Oscillatory Mobilization in chronic Mechanical Neck pain at improving Neck Disability.

To compare the effects of Cervical Retraction Exercise and Facet Oscillatory Mobilization in chronic Mechanical Neck pain at Improving Range of Motion The study design used for this literature would be Randomized Control Trial This study would include total 32 participants which would be divided into two groups, 16 each.

DETAILED DESCRIPTION:
Neck pain is a common disorder in the general population leading to disability in terms of patient's physical, social and emotional well-being. Current data suggest that 22% to 70% of people experience neck pain at some point of their lives. In the developed world, the prevalence of the chronic neck pain is reported to be ranging from 7% to 22% among women and from 5% to 16% among men. Prevalence studies showed that cervical pain is more prevalent among middle-aged women compared to their male counterparts. When the duration of symptoms is greater than 12 weeks of evolution, it acquires the value of chronicity. Chronic neck pain, occurring in approximately 50% of the global population, has a substantial societal burden. Adults with neck pain commonly experience hyperalgesia of cervical muscles, as evidenced by a reduced pressure pain threshold. Neck pain incidence raises with age and is greatest in the third and fourth decades of life with more prevalence in females. The reduced range of neck motion (ROM) is another objective finding widely investigated in chronic neck pain. It could be argued that the optimal functioning of the cervical musculature is related to the ROM; changes in neck muscle activation that result in an altered stiffness distribution may affect cervical passive stability as well as the passive and active ROM. When evaluating a patient with neck pain, the physician must be alert for red flags in the history and physical examination that may indicate the need for urgent testing and intervention. NNP is a symptom with a multifactorial etiology, and studies show its strong correlation with depression, anxiety, headache, sedentary life, sleep disorders and smoking. Risk factors for developing NNP include cervical trauma such as whiplash, sports injuries and sedentary seated work(10) Musculoskeletal disorders occurring in the neck include neck pain, cervical strain, sprain, facet joint syndrome, ruptured cervical disk, and myofascial pain syndrome, common symptoms caused by these diseases include neck pain, decreased joint range of motion, and muscle over-tension. Neck pain, which is the most common in neck diseases, limits the range of motion of the neck and causes neck dysfunction by causing crepitation and stiffness of the neck. The structural arrangement of the cervical spine makes it susceptible to mechanical changes, often triggered by degenerative shifts and improper posture, resulting in prevalent neck discomfort, with a 54% prevalence rate over 6 months. There are many methods of diagnosis both radiological and manual testing. Radiological tests include X.RAY, MRI, and CT. while manual testing includes compression and traction tests to rule out neurological or joint dysfunction. Palpation to check tenderness and manual muscle testing for neck muscles strength. Physical therapy interventions for chronic neck pain include diverse treatment approaches including manual therapy, isometrics, heating modalities stretching etc. that not only reduces pain but also increases functional ability of patient. From physiotherapist point of view it's important to use an effective manual technique that provides us with highest pain relief, improve mobility and maximum functional restoration and NAGS and SNAGS by brain mulligan are an effective approach. Cervical retraction exercise is performed with patients either in sitting or standing in an upright position while pushing their chin backward and simultaneously raising their head within the pain-free range (3 seconds). In manual therapy, joints are assessed and treated relying on the current knowledge about their kinematics, however, only limited information is available about the upper cervical spine and how its kinematics are influenced by manual mobilization. In terms of preference of techniques for the management of neck pain, exercise therapy and manual therapy are mostly applied by physiotherapists. Manual therapy techniques include joint mobilization and soft tissue mobilization techniques. Restoration of joint arthrokinematics is achieved by joint mobilizations, whereas soft tissue techniques, such as muscle energy techniques (MET) and static stretching, focus on flexibility of soft tissues, like extensibility of muscle and connective tissues. Conventional static stretching is commonly applied in the management of neck pain and other mechanical disorders, but it directs effect only on the passive component of muscle, like connective tissues or perimysium, whereas METs focus on the active component of muscle tone in addition to the passive component.

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.

  * Participants were patients with a complaint of Chronic Mechanical neck pain (> 6 weeks).
  * Neck Disability Index (NDI) score > 16%
  * Age between 35-50 years, Both Male and Female
  * NPRS score >3-6.
  * Recurrent neck pain aggravated at least once in the month.
  * Painful Cervical ROM (Flexion <80 Extension<70 rotation<90 to both sides and lateral flexion <35 degree.
  * Spurling test negative
  * Patients willing to participates in the study after filling the consent form.
  * Upper Limb Nerve tension test (Median, Radial, and Ulnar negative).

Exclusion Criteria:

* Participant failing to fall in this category would be excluded of the study.

  * Cervical radiculopathy
  * Cervical canal stenosis
  * Severe neurological disorder
  * Previous cervical surgery
  * Recent history of fall/trauma to the cervical spine.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-13 (Estimated); Study Completion 2024-12-13 (Estimated)

PRIMARY OUTCOMES:
Neck disability index | 6 weeks
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
  Score: /50 Transform to percentage score x 100 = %points. It has 7 items for daily living, 2 for pain and 1 for concentration. Each item is rated from 0 to 5. Total score is presented in percentage. Higher score tells greater disability while 0 means no disability. Total score is 50. In cervical radiculopathy patients it has moderate test retest reliability ICC= 0.68 .The NDI has a fair to moderate test-retest reliability in patients with mechanical neck pain but also for patients with cervical radiculopathy. The NDI has a good construct validity.
Numerical pain rating scale | 6 weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r = 0.96 and 0.95, respectively) before and after medical consultation.
Inclinometer | 6 weeks
  An inclinometer is a device used to measure angles. It is commonly used in physiotherapy to measure the range of motion (ROM) of joints and very similar to a goniometer.
  The digital inclinometer demonstrated excellent reliability (ICC=0.75-0.86), except for the right lateral flexion (ICC=0.74) and left rotation (ICC=0.72).

CONTACTS AND LOCATIONS:
Overall Officials: Faheem Ullah Jan, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Khyber Teaching hospital, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alansari SM, Youssef EF, Shanb AA. Efficacy of manual therapy on psychological status and pain in patients with neck pain. A randomized clinical trial. Saudi Med J. 2021 Jan;42(1):82-90. doi: 10.15537/smj.2021.1.25589. PMID 33399175
- [Background] Phadke A, Bedekar N, Shyam A, Sancheti P. Effect of muscle energy technique and static stretching on pain and functional disability in patients with mechanical neck pain: A randomized controlled trial. Hong Kong Physiother J. 2016 Apr 14;35:5-11. doi: 10.1016/j.hkpj.2015.12.002. eCollection 2016 Dec. PMID 30931028